CLINICAL TRIAL: NCT02909881
Title: Dose Response Oxidation of a Sweet-corn Derived Polysaccharide (PhytoSpherix) During Exercise in Endurance Trained Athletes
Brief Title: Dose Response Oxidation of a Sweet-corn Derived Sugar (PhytoSpherix) During Exercise in Endurance Trained Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Mirexus Biotechnologies Inc (Unknown)
Responsible Party: Principal Investigator, Peter Lemon, Professor, University of Western Ontario, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10014597
Record Dates: First submitted 2016-09-10; First posted 2016-09-21 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Hypoglycemia
Keywords: polysaccharide; oxidation; endurance exercise
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endurance trained male cyclists (Experimental): 8 male endurance trained male cyclist will consume varying amounts (0, 1, 1.5 and 2 g/min) of PhytoSpherix (sweet-corn derived sugar) during a 150 min . cycling exercise
  Interventions: Dietary Supplement: Use of PhytoSpherix at 0 g/min; Dietary Supplement: Use of PhytoSpherix at 1 g/min; Dietary Supplement: Use of PhytoSpherix at 1.5 g/min; Dietary Supplement: Use of PhytoSpherix at 2 g/min; Behavioral: Cycling exercise

INTERVENTIONS:
Dietary Supplement: Use of PhytoSpherix at 0 g/min — PhytoSpherix (Sweet-corn derived sugar) will be fed at 0 g/min during a 150 min cycling exercise
Dietary Supplement: Use of PhytoSpherix at 1 g/min — PhytoSpherix (Sweet-corn derived sugar) will be fed at 1 g/min during a 150 min cycling exercise
Dietary Supplement: Use of PhytoSpherix at 1.5 g/min — PhytoSpherix (Sweet-corn derived sugar) will be fed at 1.5 g/min during a 150 min cycling exercise
Dietary Supplement: Use of PhytoSpherix at 2 g/min — PhytoSpherix (Sweet-corn derived sugar) will be fed at 2 g/min during a 150 min cycling exercise
Behavioral: Cycling exercise — Male endurance athletes will complete a cycling exercise for 150 min at 50% of their respective maximum wattage

SUMMARY:
PhytoSpherix (Phx) is an all-natural, edible polysaccharide extracted from sweet corn. This carbohydrate is the major muscle fuel for intense exercise and its stores are quite small such that one can run out of it during a single exercise bout. Therefore, Phx should provide significant exercise fuel if consumed during exercise. As a result its intake could enhance intense exercise performance by providing additional fuel. This experiment Will investigate the effects of 4 different dosages of Phx consumed throughout a prolonged exercise bout on carbohydrate and fat utilization as well as its oxidation rate and perception of effort during prolonged intense exercise in trained cyclists. Muscle and liver carbohydrate stores will be examined using a non-invasive ultrasound technique.

DETAILED DESCRIPTION:
Carbohydrate (CHO) is one of the main substrate oxidized during moderate-to-high intensity, endurance-type exercise. It's been shown that CHO feeding during exercise enhances endurance performance and capacity, attributed mainly to the facilitation of greater rates of exogenous CHO oxidation, prevention of hypoglycaemia and sparing of muscle glycogen. Previous studies based on supplementation of glucose during 180 min. of cycling exercise have reported a maximal rate of exogenous CHO oxidation to be about 1 g/min. Other studies have shown that CHO oxidation rates can reach peak values of about 1.3 g/min when a combination of fructose and glucose is ingested at a rate of 1.8 g/min. The limitation in uptake and oxidation of a single CHO source is attributed to its intestinal transporter saturation such that when multiple CHO source is used the uptake and oxidation rate is increased to a greater extent. Currently there is no information regarding Phx uptake or oxidation rate as a CHO source during exercise. Also, it is important to investigate whether Phx as a CHO sport drink can increase performance by sparing muscle and liver glycogen during exercise. Therefore, the objective of this experiment is to measure dose response of Phx oxidation rate during prolonged cycling exercise and its effect on muscle and liver glycogen levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male endurance trained athletes with >2 y cycling experience; about 2 h/day

Exclusion Criteria:

* Unhealthy athletes, smokers

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Oxidation of PhytoSpherixat | 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session
  Breath samples will be taken starting at 0, 15, 30, 45, 60, 75, 90, 135, up to 150 min from the beginning of the exercise session to measure change in oxidation of PhytoSpherix
Noninvasive ultrasound measure of glycogen in Vastus lateralis, rectus femoris and liver | 10 min before and 10 min after the 150 min exercise session
  Change in muscle and liver glycogen will be measured 10 min before and 10 min after exercise session. When muscle and liver glycogen content is high, the ultrasound image is hypoechoic (dark), and with glycogen depletion and water loss, the image is hyperchoic (brighter).Three ultrasound measurements at each site will be made by a trained technician using a 12 MHz linear transducer and a standard diagnostic high resolution GE LOGIQ-e ultrasound machine (GE Healthcare, Milwaukee, WI). After calculating statistics on the color bar to determine the general brightness settings of the machine, images will be pre-processed and segmented to isolate the muscle area under analysis using a center crop within the muscle section 25 mm from the top muscle sheath. Comparing these results will help better understand the effect of supplementation of Phx at different rates on any changes in glycogen stores of muscle and liver.

SECONDARY OUTCOMES:
blood glucose concentration | 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session
  Changes in blood glucose will be measured at 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session. A blood drop by finger prick approach starting at time 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session under sterile practice will be used to determine blood glucose concentrations
blood lactate concentration | 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session
  Changes in blood lactate will be measured at 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session. A blood drop by finger prick approach starting at time 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session under sterile practice will be used to determine blood lactate concentrations
Respiratory exchange ratio | At 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session
  Respiratory exchange ratio will be measured at 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session for periods of 4 min by using an online automated gas-analysis system.
rate of perceived exertion | At 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session
  rate of perceived exertion (RPE) for whole body and legs will be measured at 0, 15, 30, 45, 60, 75, 90, 135, 150 min from the beginning of the exercise session on a scale from 6 to 20, using the Borg category scale.
questionnaire to rate possible gastrointestinal (GI) problems | At 30, 60, 90, 120 and 150 min from the beginning of the exercise session
  every athlete will be asked at 30, 60, 90, 120 and 150 min from the beginning of the exercise session to fill in a questionnaire to rate possible gastrointestinal (GI) problems including stomach problems, GI cramping, bloated feeling, diarrhea, nausea, dizziness, headache, belching, vomiting, and urge to urinate and defecate. While cyclists are on the bike and continue their exercise, each question will be answered by simply ticking a box on the questionnaire that corresponds to the severity of the GI problem addressed. The items will be scored on a 10-point scale (1 not at all, 10 very, very much).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Research Laboratory, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bandegan A, Huang L, Longstaffe FJ, Lemon PW. Dose-Response Oxidation of Ingested Phytoglycogen during Exercise in Endurance-Trained Men. J Nutr. 2021 Oct 1;151(10):2942-2948. doi: 10.1093/jn/nxab219. PMID 34255078